CLINICAL TRIAL: NCT02697500
Title: Pre-analytical Sample Handling Conditions and Their Effects on the Human Serum Metabolome
Status: Completed | Type: Observational
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Baer, Supervisory Research Physiologist, USDA Beltsville Human Nutrition Research Center
Other Study IDs: HS53
Record Dates: First submitted 2016-02-12; First posted 2016-03-03 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — serum and urine
Oversight: Data Monitoring Committee: No

SUMMARY:
This study evaluates how blood serum handling conditions can affect the concentrations of ~1,000 serum metabolites and attempts to quantify the degree of attenuation and/or potential bias in epidemiologic associations that may result from less than optimal sample handling conditions.

DETAILED DESCRIPTION:
Metabolomics, the simultaneous quantification of concentrations of hundreds or thousands of metabolites simultaneously in a biological matrix, is a versatile analytical technique capable of accelerating biomarker-based discoveries in nutritional science. Recently, metabolomics has been applied to samples collected in feeding studies (1) and epidemiologic studies (2) to identify dozens of novel potential dietary biomarkers. Several large prospective cohort studies, many of which are collaborating in a metabolomics consortium led by the National Cancer Institute, have recently applied metabolomics to banked samples. This has made nutrition-related biomarkers suddenly available for tens of thousands of participants with follow-up for disease endpoints, enabling truly large-scale nutritional biomarkers and disease studies.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 65 years at beginning of study.
* BMI between 18.5 and 35.0 kg/m2.

Exclusion Criteria:

* Presence of cardiovascular disease, kidney disease, liver disease, gout, hyperthyroidism, untreated or unstable hypothyroidism, certain cancers, gastrointestinal disease, pancreatic disease, other metabolic diseases, or malabsorption syndromes.
* Unable or unwilling to give informed consent or communicate with study staff.
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women will be recruited from the area surrounding the BHNRC. There are several thousand government and privately employed workers located within a 10-mile radius of the BHNRC and several residential communities from which a cohort of volunteers will be recruited. The population includes an ethnically diverse group of subjects.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2016-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Selected intensity of biochemicals identified from liquid and gas chromatography with mass ranging from 50 to 800 molecular weight. | on day one
  Serum metabolomics profiling will be conducted at Metabolon, Inc. after the serum has been handled in a number of different ways (refrigerated for different lengths of time and frozen and thawed various numbers of times)

CONTACTS AND LOCATIONS:
Locations (1):
- USDA-ARS, Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States